CLINICAL TRIAL: NCT00998023
Title: Patient Comfort Study With Vascular Closure: Mynx vs. Angio-Seal Evolution
Brief Title: Patient Comfort With Vascular Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Access Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 479-2009
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Results first posted 2011-12-06 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-11

CONDITIONS: Vascular Closure
Keywords: Angiogram; Catheter Angiogram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mynx VCD (Experimental): Mynx Vascular Closure Device
  Interventions: Device: Mynx Vascular Closure Device
- AngioSeal VCD (Active Comparator): AngioSeal Vascular Closure Device
  Interventions: Device: AngioSeal Vascular Closure Device

INTERVENTIONS:
Device: Mynx Vascular Closure Device — Comparison of two different vascular closure devices.
  Other Names: Mynx
  Arms: Mynx VCD
Device: AngioSeal Vascular Closure Device — Comparison of two different vascular closure devices.
  Other Names: AngioSeal
  Arms: AngioSeal VCD

SUMMARY:
The purpose of this research study is to collect information on the amount of discomfort patients experience with one of two different vascular blood vessel closure devices, the MynxM5 Vascular Closure Device and the Angio-Seal Evolution Vascular Closure Device.

DETAILED DESCRIPTION:
The traditional, standard technique of achieving femoral artery hemostasis following diagnostic and interventional catheterization procedures requires compression methods such as manual pressure or clamps held at the puncture site for 10 to 30 minutes, or even longer depending on sheath size and anticoagulation status. This traditional method can be associated with patient discomfort as well as prolonged bed rest, ambulation and hospital discharge.

Over the past decade, Vascular Closure Devices (VCDs), which include collagen hemostasis devices, percutaneous suture-mediated closure devices and metallic clips, have emerged as a novel means for reducing time to hemostasis and ambulation following catheterization procedures performed utilizing femoral arterial access. Previous studies with commercially available VCDs have shown that the reduction in time to hemostasis and time to ambulation and discharge have also led to increased patient satisfaction over manual compression.

The MynxM5 Vascular Closure Device received FDA approval on April 8, 2009. Like the Mynx 6/7F Vascular Closure Device, which received FDA approval on May 16, 2007, both are designed to achieve femoral artery hemostasis via delivery of an extravascular, water-soluble synthetic sealant which expands upon contact with subcutaneous fluids to seal the arteriotomy. In theory, the lack of pressure needed to clamp, suture, clip or cinch, which is required with intravascular closure devices, may provide an advantage in regards to increased patient comfort during closure device deployment when using the Mynx.

Although VCDs have demonstrated an increase in patient comfort and satisfaction over manual compression, little data exists regarding patient comfort when comparing different closure devices. This study is designed to evaluate patient comfort between the MynxM5 and Angio-Seal Evolution Vascular Closure Devices.

ELIGIBILITY:
Inclusion Criteria:

* Patient is >18 years of age
* Patient has been informed and understands the nature of the study and provides written Informed Consent approved by the appropriate Institutional Review Board prior to enrollment
* Patient has been trained and understands the use of the 0-10 Visual Analogue Scale as an assessment of patient pain
* Patient is scheduled to undergo a diagnostic endovascular procedure involving percutaneous access through the common femoral artery

Exclusion Criteria:

* Per Mynx and Angio-Seal Instructions for Use
* Patient has a documented psychiatric disorder (e.g. major depression, anxiety)
* Patient has a documented chronic pain condition requiring daily treatment
* Patient carries the diagnoses of a known bleeding disorder
* Intraprocedural Exclusion Criteria: Patient has a baseline ipsilateral groin pain rating of >1 on the 0-10 Visual Analog Scale prior to closure device deployment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Mocco, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the clinical practice of the investigator between November 2009 and July 2010.
Pre-assignment Details: Participants who had any groin pain before placement of the closure device were excluded.
Period: Overall Study
Arm/Group | Mynx VCD | AngioSeal VCD
Started | 32 | 32
Completed | 32 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mynx VCD | AngioSeal VCD | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 22 | 48
  >=65 years | 6 | 10 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 10 | 13 | 23
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Mean Score on the Visual Analogue Scale
Description: The Visual Analogue Scale measures the severity of pain on a continuous scale from 0 (no pain) to 10 (worst possible pain).
Time Frame: Immediately before vascular closure and immediately after vascular closure.
Population: Per protocol
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Mynx VCD | AngioSeal VCD
Number analyzed (Participants) | 32 | 32
Scores on a Scale
  Before Closure | 0.63 (1.01) | 0.59 (1.04)
  After Closure | 2.94 (0.42) | 5.03 (0.56)

2. Secondary Outcome: Major Complications
Description: Number of participants with permanent access site-related nerve injury, access-site related surgical/vascular repair, amputation related to access closure complication, access site-related bleeding/hematoma requiring transfusion, any new ipsilateral lower extremity ischemia requiring non-surgical intervention, local access site-related or generalized infection requiring prolonged hospitalization or re-hospitalization and treatment with IV antibiotics or inflammatory reaction that may include local signs and drainage, treated with re-hospitalization, IV antibiotics and/or surgical intervention
Time Frame: 1 Day
Population: Per protocol
Measure: Number; unit: Participants
Arm/Group | Mynx VCD | AngioSeal VCD
Number analyzed (Participants) | 32 | 32
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Mynx VCD | AngioSeal VCD
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

LIMITATIONS AND CAVEATS:
The Angio-Seal Evolution is only one of a variety of potential vascular closure devices available on the market that would be suitable for comparison with the Mynx; however, this study was limited to just one of such alternative devices.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes